CLINICAL TRIAL: NCT02422615
Title: A Randomized Double-blind, Placebo-controlled Study of Ribociclib in Combination With Fulvestrant for the Treatment of Men and Postmenopausal Women With Hormone Receptor Positive, HER2-negative, Advanced Breast Cancer Who Have Received no or Only One Line of Prior Endocrine Treatment
Brief Title: Study of Efficacy and Safety of LEE011 in Men and Postmenopausal Women With Advanced Breast Cancer.
Acronym: MONALEESA-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLEE011F2301; 2015-000617-43 (EudraCT Number)
Record Dates: First submitted 2015-04-01; First posted 2015-04-21 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Advanced Breast Cancer
Keywords: HR-positive; HER2-negative; Advanced breast cancer; LEE011; ribociclib; fulvestrant; faslodex; CDK; CDK4; CDK6; CDK4/6; CDK4/6 inhibitor; Phase III; ER-positive; PR-positive; Postmenopausal; Men; Breast Neoplasms; Breast Diseases; Neoplasms; Neoplasms by Site; Antineoplastic Agents; Antineoplastic Agents, Hormonal; Estrogen Receptor Antagonists; Hormone Antagonists; Hormones, Hormone Substitutes, and Hormone Antagonists; Molecular Mechanisms of Pharmacological Action; Pharmacologic Actions; Therapeutic Use
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Breast Neoplasms; Breast Diseases; Neoplasms; Neoplasms by Site | interventions — ribociclib; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Following protocol amendment 4 (29-Jan-2020), study participants were unblinded, with an opportunity for those patients still in the study in the arm of placebo + fulvestrant to transition to the treatment of ribociclib + fulvestrant.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ribociclib + fulvestrant (Experimental): Ribociclib was administered orally at a daily dose of 600mg for 21 consecutive days within a 28-day cycle. This treatment was combined with fulvestrant, which was administered via intramuscular injections of 500mg every 28 days starting on Day 1 of each cycle. Additionally, an extra dose of fulvestrant was given on Day 15 of Cycle 1. For participants who did not tolerate the protocol-specified dosing schedule, dose adjustments were permitted in order to allow the patient to continue the study treatment.
  Interventions: Drug: Ribociclib; Drug: Fulvestrant
- Placebo + fulvestrant (Placebo Comparator): Placebo was administered orally for 21 consecutive days within a 28-day cycle. This treatment was combined with fulvestrant, which was administered via intramuscular injections of 500mg every 28 days starting on Day 1 of each cycle. Additionally, an extra dose of fulvestrant was given on Day 15 of Cycle 1. For participants who did not tolerate the protocol-specified dosing schedule, dose adjustments were permitted in order to allow the patient to continue the study treatment.
  Participants were unblinded after the implementation of protocol amendment 4 (29-Jan-20) and were given the option to crossover to treatment with ribociclib and fulvestrant.
  Interventions: Drug: Fulvestrant; Drug: Placebo

INTERVENTIONS:
Drug: Ribociclib — Ribociclib capsules were administered orally at a daily dose of 600mg for 21 consecutive days within a 28-day cycle.
  Other Names: LEE011
  Arms: Ribociclib + fulvestrant
Drug: Fulvestrant — Fulvestrant was administered via intramuscular injections at a dose of 500mg every 28 days, starting on Day 1 of each cycle. In Cycle 1, an additional dose of Fulvestrant was given on Day 15.
Drug: Placebo — Placebo capsules were administered orally for 21 consecutive days within a 28-day cycle.
  Arms: Placebo + fulvestrant

SUMMARY:
The main aim of this study was to evaluate the efficacy and safety of adding ribociclib to fulvestrant in men and postmenopausal women with hormone receptor positive (HR+), HER2-negative advanced breast cancer.

DETAILED DESCRIPTION:
This study was a randomized, phase III, double-blind, placebo-controlled international trial aimed at determining the efficacy and safety of treatment with fulvestrant in combination with ribociclib compared to fulvestrant with placebo in men and postmenopausal women diagnosed with HR+, HER2-negative advanced breast cancer. The study comprised four phases: screening (up to 28 days), randomized treatment, post-treatment disease progression follow-up, and post-treatment survival follow-up.

Enrolled participants were randomly assigned to receive either fulvestrant+ribociclib or fulvestrant+placebo in a ratio of 2:1. The randomization process was stratified based on the presence of liver and/or lung metastases (yes versus no) and prior endocrine therapy. Treatment was administered until disease progression, occurrence of unacceptable toxicity, or discontinuation from the study treatment for other reasons.

Participants who discontinued treatment due to reasons other than disease progression or withdrawal of consent for efficacy follow-up continued to be monitored until disease progression, death, withdrawal of consent, loss to follow-up, or subject/guardian decision.

All participants who discontinued treatment were followed for survival until the predetermined number of overall survival (OS) events was reached.

A protocol amendment 4 (dated 29-Jan-2020) allowed for unblinding of study participants, and those still receiving placebo had the option to switch to the ribociclib arm. The decision for crossover was made at the investigator's discretion and required patient consent.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients were adults, both male and female, aged ≥ 18 years at the time of providing informed consent. Female patients were required to be postmenopausal. Informed consent was obtained prior to any trial-related activities, following local guidelines.
2. Patients had a confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer, determined through histological and/or cytological examination by a local laboratory. Patients also had HER2-negative breast cancer.
3. Patients had either measurable disease as per RECIST 1.1 criteria or at least one predominantly lytic bone lesion.
4. Patients had advanced breast cancer, which included locoregionally recurrent disease not amenable to curative therapies (such as surgery or radiotherapy) or metastatic breast cancer. Patients fell into one of the following categories:

   * Newly diagnosed with advanced/metastatic breast cancer and treatment-naïve.
   * Relapsed with documented evidence of relapse more than 12 months after completing (neo)adjuvant endocrine therapy, without any prior treatment for advanced/metastatic disease.
   * Relapsed with documented evidence of relapse on or within 12 months from completing (neo)adjuvant endocrine therapy, without any prior treatment for advanced/metastatic disease.
   * Relapsed with documented evidence of relapse more than 12 months after completing adjuvant endocrine therapy and subsequently progressed after receiving one line of endocrine therapy (antiestrogen or aromatase inhibitor) for advanced/metastatic disease.
   * Newly diagnosed with advanced/metastatic breast cancer at diagnosis and progressed after receiving one line of endocrine therapy (antiestrogen or aromatase inhibitor), with documented evidence of progression.
5. Patients had an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Patients had adequate bone marrow and organ function.

Key Exclusion Criteria:

Patients with symptomatic visceral disease or disease burden that rendered them ineligible for endocrine therapy, based on the investigator's judgment.

2. Patients who had received prior treatment with chemotherapy (except for neoadjuvant/adjuvant chemotherapy), fulvestrant, or any CDK4/6 inhibitor.

3. Patients with inflammatory breast cancer at the screening stage. 4. Patients with central nervous system (CNS) involvement, unless they were at least 4 weeks from completing prior therapy before initiating the study treatment and had a stable CNS tumor at the time of screening. They were also required not to be receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases.

5. Patients with clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality.

6. Patients who were currently receiving any of the following substances, which could not be discontinued 7 days prior to initiating treatment:

* Known strong inducers or inhibitors of CYP3A4/5.
* Substances with a known risk of prolonging the QT interval or inducing Torsades de Pointes.
* Substances with a narrow therapeutic window and predominantly metabolized through CYP3A4/5.
* Herbal preparations/medications, dietary supplements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2023-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (159):
- United States (26):
  - Southern Cancer Center PC SC-2, Mobile, Alabama
  - Ironwood Cancer and Research Centers SC-2, Chandler, Arizona
  - Highlands Oncology Group ., Fayetteville, Arkansas
  - UCLA Medical Center ., Los Angeles, California
  - Central Coast Medical Oncology Corporation SC, Santa Maria, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Florida Cancer Research Institute Dept of Oncology, Davie, Florida
  - Florida Hospital Cancer Institute SC, Orlando, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - John D Archbold Memorial Hospital Main, Thomasville, Georgia
  - Moanalua Medical Center. Attn: Oncology Dept SC, Honolulu, Hawaii
  - Oncology Specialists, SC Advocate Medical Group-Niles, Park Ridge, Illinois
  - Jackson Oncology Associates SC, Jackson, Mississippi
  - Meridian Health Systems Regulatory, Neptune City, New Jersey
  - University of New Mexico Cancer Center SC, Albuquerque, New Mexico
  - CR Wood Cancer Center SC, Glens Falls, New York
  - Clinical Research Alliance ., Lake Success, New York
  - NYU Langone Med Center CV Research NYU Langone Medical Center, New York, New York
  - Genesis Cancer Services SC, Zanesville, Ohio
  - Penn State University Milton S Hershey Medical Center SC, Hershey, Pennsylvania
  - Millennium Research Clin Develop SC, Houston, Texas
  - Northern Utah Cancer Associates CFTY720DUS01, Ogden, Utah
  - Providence Regional Cancer Partnership ., Everett, Washington
  - Providence Regional Cancer System SC, Lacey, Washington
  - Virginia Mason Medical Center-Oncology SC, Seattle, Washington
- Australia (4):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, East Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Austria (2):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Vienna
- Belgium (6):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Namur
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (12):
  - Novartis Investigative Site, Surrey, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Rimouski, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Colombia (2):
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Montería
- Czechia (4):
  - Novartis Investigative Site, Brno-Bohunice, Czech Republic
  - Novartis Investigative Site, Liberec, Czech Republic
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
- Denmark (6):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Odense C
  - Novartis Investigative Site, Vejle
- France (13):
  - Novartis Investigative Site, Strasbourg, Cedex
  - Novartis Investigative Site, Saint-Cloud, Hauts De Seine
  - Novartis Investigative Site, Reims, Marne
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Toulon La Seyne Sur Mer
- Germany (23):
  - Novartis Investigative Site, Langen, Hesse
  - Novartis Investigative Site, Georgsmarienhütte, Lower Saxony
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Fürth
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mühlhausen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Ravensburg
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Troisdorf
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Velbert
  - Novartis Investigative Site, Weiden
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szolnok
- Italy (8):
  - Novartis Investigative Site, L’Aquila, AQ
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Lecce, LE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Pontedera, PI
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Amman, Jordan
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
- Malaysia (2):
  - Novartis Investigative Site, Johor Bahru, Johor
  - Novartis Investigative Site, Kuching, Sarawak
- Novartis Investigative Site, Oaxaca City, Mexico
- Netherlands (12):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Enschede
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Hoofddorp
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Nieuwegein
  - Novartis Investigative Site, Roermond
  - Novartis Investigative Site, Sittard-Geleen
  - Novartis Investigative Site, The Hague
  - Novartis Investigative Site, Tilburg
- Novartis Investigative Site, Oslo, Norway
- Poland (2):
  - Novartis Investigative Site, Konin
  - Novartis Investigative Site, Warsaw
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Russia (2):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Tambov
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (11):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Madrid, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Sant Joan Despí, Barcelona
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, San Sebastián de los Reyes, Madrid
  - Novartis Investigative Site, Madrid
- Sweden (3):
  - Novartis Investigative Site, Eskilstuna
  - Novartis Investigative Site, Sundsvall
  - Novartis Investigative Site, Vaxjo
- Switzerland (3):
  - Novartis Investigative Site, Aarau
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Zurich
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- United Kingdom (2):
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Hart LL, Im SA, Tolaney SM, Campone M, Pluard T, Sousa B, Freyer G, Decker T, Kalinsky K, Sopher G, Gao M, Hu H, Kuemmel S. Efficacy, safety, and patient-reported outcomes across young to older age groups of patients with HR+/HER2- advanced breast cancer treated with ribociclib plus endocrine therapy in the randomized MONALEESA-2, -3, and -7 trials. Eur J Cancer. 2025 Feb 25;217:115225. doi: 10.1016/j.ejca.2025.115225. Epub 2025 Jan 8. PMID 39826197
- [Derived] Andre F, Su F, Solovieff N, Hortobagyi G, Chia S, Neven P, Bardia A, Tripathy D, Lu YS, Lteif A, Taran T, Babbar N, Slamon D, Arteaga CL. Pooled ctDNA analysis of MONALEESA phase III advanced breast cancer trials. Ann Oncol. 2023 Nov;34(11):1003-1014. doi: 10.1016/j.annonc.2023.08.011. Epub 2023 Sep 5. PMID 37673211
- [Derived] Neven P, Fasching PA, Chia S, Jerusalem G, De Laurentiis M, Im SA, Petrakova K, Bianchi GV, Martin M, Nusch A, Sonke GS, De la Cruz-Merino L, Beck JT, Zarate JP, Wang Y, Chakravartty A, Wang C, Slamon DJ. Updated overall survival from the MONALEESA-3 trial in postmenopausal women with HR+/HER2- advanced breast cancer receiving first-line ribociclib plus fulvestrant. Breast Cancer Res. 2023 Aug 31;25(1):103. doi: 10.1186/s13058-023-01701-9. PMID 37653397
- [Derived] Ji Y, Yartsev V, Quinlan M, Serra P, Wang Y, Chakraborty A, Miller M. Justifying Ribociclib Dose in Patients with Advanced Breast Cancer with Renal Impairment Based on PK, Safety, and Efficacy Data: An Innovative Approach Integrating Data from a Dedicated Renal Impairment Study and Oncology Clinical Trials. Clin Pharmacokinet. 2023 Mar;62(3):493-504. doi: 10.1007/s40262-022-01206-2. Epub 2023 Feb 17. PMID 36800111
- [Derived] Burris HA, Chan A, Bardia A, Thaddeus Beck J, Sohn J, Neven P, Tripathy D, Im SA, Chia S, Esteva FJ, Hart L, Zarate JP, Ridolfi A, Lorenc KR, Yardley DA. Safety and impact of dose reductions on efficacy in the randomised MONALEESA-2, -3 and -7 trials in hormone receptor-positive, HER2-negative advanced breast cancer. Br J Cancer. 2021 Aug;125(5):679-686. doi: 10.1038/s41416-021-01415-9. Epub 2021 Jun 22. PMID 34158598
- [Derived] Slamon DJ, Neven P, Chia S, Jerusalem G, De Laurentiis M, Im S, Petrakova K, Valeria Bianchi G, Martin M, Nusch A, Sonke GS, De la Cruz-Merino L, Beck JT, Ji Y, Wang C, Deore U, Chakravartty A, Zarate JP, Taran T, Fasching PA. Ribociclib plus fulvestrant for postmenopausal women with hormone receptor-positive, human epidermal growth factor receptor 2-negative advanced breast cancer in the phase III randomized MONALEESA-3 trial: updated overall survival. Ann Oncol. 2021 Aug;32(8):1015-1024. doi: 10.1016/j.annonc.2021.05.353. Epub 2021 Jun 5. PMID 34102253
- [Derived] Prat A, Chaudhury A, Solovieff N, Pare L, Martinez D, Chic N, Martinez-Saez O, Braso-Maristany F, Lteif A, Taran T, Babbar N, Su F. Correlative Biomarker Analysis of Intrinsic Subtypes and Efficacy Across the MONALEESA Phase III Studies. J Clin Oncol. 2021 May 1;39(13):1458-1467. doi: 10.1200/JCO.20.02977. Epub 2021 Mar 26. PMID 33769862
- [Derived] Slamon DJ, Neven P, Chia S, Fasching PA, De Laurentiis M, Im SA, Petrakova K, Bianchi GV, Esteva FJ, Martin M, Nusch A, Sonke GS, De la Cruz-Merino L, Beck JT, Pivot X, Sondhi M, Wang Y, Chakravartty A, Rodriguez-Lorenc K, Taran T, Jerusalem G. Overall Survival with Ribociclib plus Fulvestrant in Advanced Breast Cancer. N Engl J Med. 2020 Feb 6;382(6):514-524. doi: 10.1056/NEJMoa1911149. Epub 2019 Dec 11. PMID 31826360
- [Derived] Yardley DA. MONALEESA clinical program: a review of ribociclib use in different clinical settings. Future Oncol. 2019 Aug;15(23):2673-2686. doi: 10.2217/fon-2019-0130. Epub 2019 Jul 15. PMID 31305131
- [Derived] Slamon DJ, Neven P, Chia S, Fasching PA, De Laurentiis M, Im SA, Petrakova K, Bianchi GV, Esteva FJ, Martin M, Nusch A, Sonke GS, De la Cruz-Merino L, Beck JT, Pivot X, Vidam G, Wang Y, Rodriguez Lorenc K, Miller M, Taran T, Jerusalem G. Phase III Randomized Study of Ribociclib and Fulvestrant in Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: MONALEESA-3. J Clin Oncol. 2018 Aug 20;36(24):2465-2472. doi: 10.1200/JCO.2018.78.9909. Epub 2018 Jun 3. PMID 29860922

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 174 sites across 30 countries enrolled participants
Pre-assignment Details: Screening assessments were conducted up to 28 days prior to the randomization
Groups:
- Ribociclib + Fulvestrant: Ribociclib was administered orally at a daily dose of 600mg for 21 consecutive days within a 28-day cycle. This treatment was combined with fulvestrant, which was administered via intramuscular injections of 500mg every 28 days starting on Day 1 of each cycle. Additionally, an extra dose of fulvestrant was given on Day 15 of Cycle 1.
- Placebo + Fulvestrant: Placebo was administered orally for 21 consecutive days within a 28-day cycle. This treatment was combined with fulvestrant, which was administered via intramuscular injections of 500mg every 28 days starting on Day 1 of each cycle. Additionally, an extra dose of fulvestrant was given on Day 15 of Cycle 1. Participants were unblinded after the implementation of protocol amendment 4 (29-Jan-20) and were given the option to crossover to treatment with ribociclib and fulvestrant.
Period: Treatment Period
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant
Started | 484 | 242
Untreated | 1 | 1
Crossover Cohort (Participants in the placebo+fulvestrant arm who crossed over to the ribociclib+fulvestrant arm and received at least one dose of the study treatment.) | 0 | 3
Completed (Treatment ongoing at the time of the cut-off 11-Jan-2023) | 0 | 0
Not Completed | 484 | 242
Not completed — Progressive disease | 314 | 200
Not completed — Adverse Event | 51 | 9
Not completed — Physician Decision | 32 | 8
Not completed — Subject/guardian decision | 38 | 8
Not completed — Death | 2 | 1
Not completed — Technical problems | 0 | 1
Not completed — Protocol deviation | 1 | 1
Not completed — Study terminated as per protocol | 46 | 14
Period: Post-treatment Efficacy Follow-up
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant
Started | 34 | 9
Completed | 0 | 0
Not Completed | 34 | 9
Not completed — Adverse Event | 1 | 0
Not completed — Death | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Progressive disease | 23 | 6
Not completed — Study Terminated as per protocol | 2 | 0
Not completed — Subject/Guardian Decision | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant | Total
Number analyzed (Participants) | 484 | 242 | 726
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (9.78) | 62.8 (10.59) | 63.2 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 484 | 242 | 726
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 406 | 213 | 619
  Asian | 45 | 18 | 63
  Native American | 5 | 1 | 6
  Black | 3 | 2 | 5
  Other | 10 | 3 | 13
  Unkown | 15 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Per Investigator Assessment
Description: PFS was defined as the period starting from the date of randomization to the date of the first documented progression or death caused by any reason. In cases where patients did not experience an event, the PFS was censored at the date of the last adequate tumor assessment. Clinical deterioration without objective radiological evidence was not considered as documented disease progression.
  PFS was assessed via local radiology assessment according to RECIST 1.1. The Kaplan-Meier method was used to estimate PFS, and the median PFS, along with 95% confidence intervals, was reported for each treatment group.
  The distribution of PFS between the two arms was compared using a stratified log-rank test at a one-sided 2.5% level of significance. The PFS hazard ratio with two-sided 95% confidence interval was derived from the stratified Cox proportional hazards model.
Time Frame: From randomization to first documented progression or death, assessed up to approximately 26 months
Population: The Full Analysis Set (FAS) including all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Placebo + Fulvestrant: Placebo was administered orally for 21 consecutive days within a 28-day cycle. This treatment was combined with fulvestrant, which was administered via intramuscular injections of 500mg every 28 days starting on Day 1 of each cycle. Additionally, an extra dose of fulvestrant was given on Day 15 of Cycle 1.
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 484 | 242
Months | 20.5 [18.5 to 23.5] | 12.8 [10.9 to 16.3]
Statistical Analysis 1: Comparison: Ribociclib + Fulvestrant vs Placebo + Fulvestrant; Test type: Superiority; p = 0.00000041, Log Rank; Cox Proportional Hazard = 0.593, 95% CI 2-sided [0.480 to 0.732]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause. In cases where the patient's death was not recorded, the OS value was censored at the date of the last known patient's survival status. As per protocol, the final OS analysis was conducted after approximately 351 deaths were documented.
  OS was estimated using the Kaplan-Meier method. The median OS, along with 95% confidence intervals (CIs), was reported for each treatment group.
  The distribution of OS between the two treatment arms was compared using a log-rank test at one-sided cumulative 2.5% level of significance. A stratified Cox regression was used to estimate the OS hazard ratio and the associated 95% CI.
Time Frame: From randomization to death, assessed up to approximately 46 months
Population: FAS including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 484 | 242
Months | NA [42.5 to NA] — NA: Not estimable due to the insufficient number of participants with events | 40.0 [37.0 to NA] — NA: Not estimable due to the insufficient number of participants with events
Statistical Analysis 1: Comparison: Ribociclib + Fulvestrant vs Placebo + Fulvestrant; Test type: Superiority; p = 0.00455, Log Rank; Cox Proportional Hazard = 0.724, 95% CI 2-sided [0.568 to 0.924]

3. Secondary Outcome: Progression Free Survival (PFS) Per Blinded Independent Review Committee (BIRC)
Description: PFS was defined as the period starting from the date of randomization to the date of the first documented progression or death caused by any reason. In cases where patients did not experience an event, the PFS was censored at the date of the last adequate tumor assessment. Clinical deterioration without objective radiological evidence was not considered as documented disease progression.
  PFS was assessed via BIRC assessment according to RECIST 1.1. The Kaplan-Meier method was used to estimate PFS, and the median PFS, along with 95% confidence intervals, was reported for each treatment group.
Time Frame: From randomization to first documented progression or death, assessed up to approximately 26 months
Population: FAS including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 484 | 242
Months | NA [18.2 to NA] — NA: Not estimable due to the insufficient number of participants with events | 10.9 [3.8 to 17.2]
Statistical Analysis 1: Comparison: Ribociclib + Fulvestrant vs Placebo + Fulvestrant; Test type: Superiority; Cox Proportional Hazard = 0.492, 95% CI 2-sided [0.345 to 0.703]

4. Secondary Outcome: Overall Response Rate (ORR) Per Investigator Assessment
Description: ORR was defined as the percentage of participants with the best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1 as per investigator assessment.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 26 months
Population: FAS including all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 484 | 242
Percentage of participants | 32.4 [28.3 to 36.6] | 21.5 [16.3 to 26.7]

5. Secondary Outcome: Clinical Benefit Rate (CBR) Per Investigator Assessment
Description: CBR was defined as the percentage of participants with a best overall response of CR or PR or stable disease (SD) lasting 24 weeks or longer as defined in RECIST 1.1 as per investigator assessment.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 26 months
Population: FAS including all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 484 | 242
Percentage of participants | 70.2 [66.2 to 74.3] | 62.8 [56.7 to 68.9]

6. Secondary Outcome: Time to Response (TTR) Per Investigator Assessment
Description: TTR was defined as the time from randomization to the first documented and confirmed response (CR or PR) as defined by RECIST 1.1 per investigator assessment. The Kaplan-Meier method was used to estimate TTR, and the median TTR, along with 95% confidence intervals, was reported for each treatment group. Participants who did not achieve a confirmed response were censored at the maximum follow-up time for patients who had a PFS event (i.e. either progressed or died due to any cause) or at the date of last adequate tumor assessment otherwise.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From randomization to first response, assessed up to approximately 26 months
Population: FAS including all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 484 | 242
Months | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events

7. Secondary Outcome: Duration of Response (DOR) Per Investigator Assessment
Description: DOR was defined as the time from the first documented response (CR or PR) to the first documented progression or death due to underlying cancer as defined in RECIST 1.1 per investigator assessment. The Kaplan-Meier method was used to estimate DOR, and the median DOR, along with 95% confidence intervals, was reported for each treatment group. If a participant had not had an event, duration was censored at the date of last adequate tumor assessment.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From first documented response to progression or death, assessed up to approximately 26 months
Population: Randomized participants with confirmed CR or PR as per investigator assessment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 157 | 52
Months | NA [16.1 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [13.8 to NA] — NA: Not estimable due to the insufficient number of participants with events

8. Secondary Outcome: Time to Definitive Deterioration of Eastern Cooperative Oncology Group Performance Status (ECOG PS) in One Score Category
Description: ECOG PS categorized patients based on their ability to perform daily activities and self-care, with scores ranging from 0 to 5. A score of 0 indicated no restrictions in activity, while higher scores indicated increasing limitations. Time to definitive deterioration was defined as the time from the date of randomization to the date of the event, defined as experiencing an increase in ECOG PS by at least one category from the baseline or death. A deterioration was considered definitive if no improvements in the ECOG PS were observed at a subsequent time. The Kaplan-Meier method was used to estimate the distribution, and the median time to definitive deterioration, along with 95% confidence intervals, was reported for each treatment group. Patients receiving any further therapy prior to definitive worsening were censored at their date of last assessment prior to start of therapy. Patients that had not worsened at the data cutoff point were censored at the date of last assessment.
Time Frame: Up to approximately 26 months
Population: FAS including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 484 | 242
Months | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events

9. Secondary Outcome: Time to Definitive 10% Deterioration in the Global Health Status/Quality of Life (GHS/QoL) Scale Score of the European Organization for Research and Treatment of Cancer's Core Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 is a questionnaire that includes 5 functional scales, 3 symptom scales, a GHS/QoL scale, and 6 single items. GHS/QoL scale scores range between 0 and 100. A high score for GHS/QoL represents better functioning or QoL.
  The time to definitive 10% deterioration is defined as the time from the date of randomization to the date of event, which is defined as at least 10% relative to baseline worsening of the QoL score (without further improvement above the threshold) or death due to any cause. The Kaplan-Meier method was used to estimate the distribution, and the median time to definitive 10% deterioration, along with 95% confidence intervals, was reported for each treatment group. If a patient had not had an event, time to deterioration was censored at the date of the last adequate QoL evaluation.
Time Frame: Up to approximately 26 months
Population: FAS including all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 484 | 242
Months | NA [22.1 to NA] — NA: Not estimable due to the insufficient number of participants with events | 19.4 [16.6 to NA] — NA: Not estimable due to the insufficient number of participants with events

10. Secondary Outcome: Change From Baseline in the GHS/QoL Scale Score of the EORTC QLQ-C30
Description: The EORTC QLQ-C30 is a questionnaire that includes 5 functional scales, 3 symptom scales, a GHS/QoL scale, and 6 single items. GHS/QoL scale scores range between 0 and 100. A high score for GHS/QoL represents better functioning or QoL.
  The change from baseline in the GHS/QoL score was assessed. A positive change from baseline indicates improvement. For subjects who discontinued treatment without disease progression, post-treatment efficacy visits occurred every 8 weeks during the initial 18 months since start of treatment, followed by visits every 12 weeks until disease progression.
Time Frame: Baseline, every 8 weeks after randomization during 18 months, then every 12 weeks up to end of treatment; end of treatment; and every 8 or 12 weeks post-treatment until progression (post-treatment efficacy visits), assessed up to approximately 26 months
Population: Randomized participants with data available at the specified time points. Number analyzed refers to the number of participants with an evaluable value at the specified time point.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 361 | 169
Score on a Scale
  Cycle 3 Day 1 (Cycle= 28 days) | 4.5 (18.53) | 2.7 (17.50)
  Cycle 5 Day 1 (Cycle= 28 days): number analyzed (Participants) | 316 | 149
  Cycle 5 Day 1 (Cycle= 28 days) | 4.2 (19.97) | 3.2 (18.09)
  Cycle 7 Day 1 (Cycle= 28 days): number analyzed (Participants) | 300 | 133
  Cycle 7 Day 1 (Cycle= 28 days) | 4.9 (19.47) | 4.3 (17.30)
  Cycle 9 Day 1 (Cycle= 28 days): number analyzed (Participants) | 283 | 133
  Cycle 9 Day 1 (Cycle= 28 days) | 4.1 (19.36) | 3.3 (17.61)
  Cycle 11 Day 1 (Cycle= 28 days): number analyzed (Participants) | 251 | 116
  Cycle 11 Day 1 (Cycle= 28 days) | 4.9 (17.57) | 2.3 (18.21)
  Cycle 13 Day 1 (Cycle= 28 days): number analyzed (Participants) | 240 | 105
  Cycle 13 Day 1 (Cycle= 28 days) | 4.4 (18.53) | 1.3 (19.48)
  Cycle 15 Day 1 (Cycle= 28 days): number analyzed (Participants) | 218 | 96
  Cycle 15 Day 1 (Cycle= 28 days) | 3.6 (18.34) | 3.6 (19.86)
  Cycle 17 Day 1 (Cycle= 28 days): number analyzed (Participants) | 216 | 84
  Cycle 17 Day 1 (Cycle= 28 days) | 3.9 (20.31) | 3.4 (21.61)
  Cycle 19 Day 1 (Cycle= 28 days): number analyzed (Participants) | 185 | 82
  Cycle 19 Day 1 (Cycle= 28 days) | 3.8 (17.57) | 3.7 (18.52)
  Cycle 22 Day 1 (Cycle= 28 days): number analyzed (Participants) | 118 | 46
  Cycle 22 Day 1 (Cycle= 28 days) | 6.6 (20.78) | 4.7 (17.00)
  Cycle 25 Day 1 (Cycle= 28 days): number analyzed (Participants) | 54 | 19
  Cycle 25 Day 1 (Cycle= 28 days) | 5.7 (16.81) | 8.3 (18.22)
  Cycle 28 Day 1 (Cycle= 28 days): number analyzed (Participants) | 12 | 3
  Cycle 28 Day 1 (Cycle= 28 days) | 12.5 (16.48) | 19.4 (12.73)
  End of treatment (EOT): number analyzed (Participants) | 184 | 113
  End of treatment (EOT) | -5.2 (25.84) | -5.5 (24.54)
  Post EOT1: number analyzed (Participants) | 11 | 2
  Post EOT1 | 4.5 (21.20) | -33.3 (23.57)
  Post EOT2: number analyzed (Participants) | 7 | 2
  Post EOT2 | -4.8 (19.75) | -16.7 (23.57)
  Post EOT3: number analyzed (Participants) | 4 | 2
  Post EOT3 | 14.6 (24.88) | -16.7 (0.00)
  Post EOT4: number analyzed (Participants) | 5 | 1
  Post EOT4 | 10.0 (20.75) | -25.0
  Post EOT5: number analyzed (Participants) | 3 | 0
  Post EOT5 | 13.9 (20.97) |
  Post EOT6: number analyzed (Participants) | 3 | 0
  Post EOT6 | 22.2 (12.73) |
  Post EOT7: number analyzed (Participants) | 3 | 0
  Post EOT7 | 19.4 (20.97) |
  Post EOT8: number analyzed (Participants) | 2 | 0
  Post EOT8 | 37.5 (17.68) |
  Post EOT9: number analyzed (Participants) | 3 | 0
  Post EOT9 | 8.3 (46.40) |
  Post EOT10: number analyzed (Participants) | 1 | 0
  Post EOT10 | -8.3 |

11. Secondary Outcome: Ribociclib Plasma Concentrations
Description: Blood samples were collected to assess the concentration by time point for ribociclib. Participants were classified into the following dose groups at each timepoint: 1) ribociclib 600 mg: consisted of all participants who provided evaluable concentrations after receiving at least 10 consecutive daily ribociclib doses of 600 mg immediately prior to the blood collection without a dose change or interruption. 2) ribociclib 400 mg: consisted of all participants who provided evaluable concentrations after receiving at least 10 consecutive daily ribociclib doses of 400 mg immediately prior to the blood collection without a dose change or interruption. 3) ribociclib 200 mg: consisted of all participants who provided evaluable concentrations after receiving at least 10 consecutive daily ribociclib doses of 200 mg immediately prior to the blood collection without a dose change or interruption.
Time Frame: Cycle 1 and Cycle 2 at Day 15 pre-dose and at 2, 4, and 6 hours post-dose. Cycle=28 days
Population: All participants with at least one evaluable ribociclib concentration. Number analyzed indicated the number of participants with an evaluable ribociclib concentration at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng) / miliLiter (mL)
Arm/Group | Ribociclib + Fulvestrant
Number analyzed (Participants) | 253
nanogram (ng) / miliLiter (mL)
  Cycle 1 Day 15 predose (ribociclib 600 mg) | 627 (67.6)
  Cycle 1 Day 15 predose (ribociclib 400 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 predose (ribociclib 200 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 2 hours post-dose (ribociclib 600 mg): number analyzed (Participants) | 102
  Cycle 1 Day 15 2 hours post-dose (ribociclib 600 mg) | 1670 (52.0)
  Cycle 1 Day 15 2 hours post-dose (ribociclib 400 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 2 hours post-dose (ribociclib 200 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 4 hours post-dose (ribociclib 600 mg): number analyzed (Participants) | 107
  Cycle 1 Day 15 4 hours post-dose (ribociclib 600 mg) | 1690 (46.2)
  Cycle 1 Day 15 4 hours post-dose (ribociclib 400 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 4 hours post-dose (ribociclib 200 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 6 hours post-dose (ribociclib 600 mg): number analyzed (Participants) | 92
  Cycle 1 Day 15 6 hours post-dose (ribociclib 600 mg) | 1420 (50.9)
  Cycle 1 Day 15 6 hours post-dose (ribociclib 400 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 6 hours post-dose (ribociclib 200 mg): number analyzed (Participants) | 0
  Cycle 2 Day 15 predose (ribociclib 600 mg): number analyzed (Participants) | 177
  Cycle 2 Day 15 predose (ribociclib 600 mg) | 553 (80.7)
  Cycle 2 Day 15 predose (ribociclib 400 mg): number analyzed (Participants) | 7
  Cycle 2 Day 15 predose (ribociclib 400 mg) | 220 (81.6)
  Cycle 2 Day 15 predose (ribociclib 200 mg): number analyzed (Participants) | 0
  Cycle 2 Day 15 2 hours post-dose (ribociclib 600 mg): number analyzed (Participants) | 75
  Cycle 2 Day 15 2 hours post-dose (ribociclib 600 mg) | 1470 (80.7)
  Cycle 2 Day 15 2 hours post-dose (ribociclib 400 mg): number analyzed (Participants) | 7
  Cycle 2 Day 15 2 hours post-dose (ribociclib 400 mg) | 794 (85.0)
  Cycle 2 Day 15 2 hours post-dose (ribociclib 200 mg): number analyzed (Participants) | 1
  Cycle 2 Day 15 2 hours post-dose (ribociclib 200 mg) | 104
  Cycle 2 Day 15 4 hours post-dose (ribociclib 600 mg): number analyzed (Participants) | 79
  Cycle 2 Day 15 4 hours post-dose (ribociclib 600 mg) | 1610 (53.6)
  Cycle 2 Day 15 4 hours post-dose (ribociclib 400 mg): number analyzed (Participants) | 7
  Cycle 2 Day 15 4 hours post-dose (ribociclib 400 mg) | 913 (69.4)
  Cycle 2 Day 15 4 hours post-dose (ribociclib 200 mg): number analyzed (Participants) | 1
  Cycle 2 Day 15 4 hours post-dose (ribociclib 200 mg) | 112
  Cycle 2 Day 15 6 hours post-dose (ribociclib 600 mg): number analyzed (Participants) | 69
  Cycle 2 Day 15 6 hours post-dose (ribociclib 600 mg) | 1280 (89.6)
  Cycle 2 Day 15 6 hours post-dose (ribociclib 400 mg): number analyzed (Participants) | 5
  Cycle 2 Day 15 6 hours post-dose (ribociclib 400 mg) | 710 (47.4)
  Cycle 2 Day 15 6 hours post-dose (ribociclib 200 mg): number analyzed (Participants) | 1
  Cycle 2 Day 15 6 hours post-dose (ribociclib 200 mg) | 104

12. Secondary Outcome: LEQ803 Plasma Concentrations
Description: Blood samples were collected to assess the concentration by time point for LEQ803, a metabolite of ribociclib. Participants were classified into the following dose groups at each timepoint: 1) ribociclib 600 mg: consisted of all participants who provided evaluable concentrations after receiving at least 10 consecutive daily ribociclib doses of 600 mg immediately prior to the blood collection without a dose change or interruption. 2) ribociclib 400 mg: consisted of all participants who provided evaluable concentrations after receiving at least 10 consecutive daily ribociclib doses of 400 mg immediately prior to the blood collection without a dose change or interruption. 3) ribociclib 200 mg: consisted of all participants who provided evaluable concentrations after receiving at least 10 consecutive daily ribociclib doses of 200 mg immediately prior to the blood collection without a dose change or interruption.
Time Frame: Cycle 1 and Cycle 2 at Day 15 pre-dose and at 2, 4, and 6 hours post-dose. Cycle = 28 days
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ribociclib + Fulvestrant
Number analyzed (Participants) | 253
ng/mL
  Cycle 1 Day 15 predose (ribociclib 600 mg) | 75.6 (50.4)
  Cycle 1 Day 15 predose (ribociclib 400 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 predose (ribociclib 200 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 2 hours post-dose (ribociclib 600 mg): number analyzed (Participants) | 102
  Cycle 1 Day 15 2 hours post-dose (ribociclib 600 mg) | 134 (44.5)
  Cycle 1 Day 15 2 hours post-dose (ribociclib 400 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 2 hours post-dose (ribociclib 200 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 4 hours post-dose (ribociclib 600 mg): number analyzed (Participants) | 107
  Cycle 1 Day 15 4 hours post-dose (ribociclib 600 mg) | 137 (42.0)
  Cycle 1 Day 15 4 hours post-dose (ribociclib 400 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 4 hours post-dose (ribociclib 200 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 6 hours post-dose (ribociclib 600 mg): number analyzed (Participants) | 92
  Cycle 1 Day 15 6 hours post-dose (ribociclib 600 mg) | 128 (42.4)
  Cycle 1 Day 15 6 hours post-dose (ribociclib 400 mg): number analyzed (Participants) | 0
  Cycle 1 Day 15 6 hours post-dose (ribociclib 200 mg): number analyzed (Participants) | 0
  Cycle 2 Day 15 predose (ribociclib 600 mg): number analyzed (Participants) | 177
  Cycle 2 Day 15 predose (ribociclib 600 mg) | 72.7 (62.9)
  Cycle 2 Day 15 predose (ribociclib 400 mg): number analyzed (Participants) | 7
  Cycle 2 Day 15 predose (ribociclib 400 mg) | 46.2 (52.3)
  Cycle 2 Day 15 predose (ribociclib 200 mg): number analyzed (Participants) | 0
  Cycle 2 Day 15 2 hours post-dose (ribociclib 600 mg): number analyzed (Participants) | 75
  Cycle 2 Day 15 2 hours post-dose (ribociclib 600 mg) | 126 (56.4)
  Cycle 2 Day 15 2 hours post-dose (ribociclib 400 mg): number analyzed (Participants) | 7
  Cycle 2 Day 15 2 hours post-dose (ribociclib 400 mg) | 70.8 (68.5)
  Cycle 2 Day 15 2 hours post-dose (ribociclib 200 mg): number analyzed (Participants) | 1
  Cycle 2 Day 15 2 hours post-dose (ribociclib 200 mg) | 36.0
  Cycle 2 Day 15 4 hours post-dose (ribociclib 600 mg): number analyzed (Participants) | 79
  Cycle 2 Day 15 4 hours post-dose (ribociclib 600 mg) | 134 (44.9)
  Cycle 2 Day 15 4 hours post-dose (ribociclib 400 mg): number analyzed (Participants) | 7
  Cycle 2 Day 15 4 hours post-dose (ribociclib 400 mg) | 79.3 (67.2)
  Cycle 2 Day 15 4 hours post-dose (ribociclib 200 mg): number analyzed (Participants) | 1
  Cycle 2 Day 15 4 hours post-dose (ribociclib 200 mg) | 41.9
  Cycle 2 Day 15 6 hours post-dose (ribociclib 600 mg): number analyzed (Participants) | 69
  Cycle 2 Day 15 6 hours post-dose (ribociclib 600 mg) | 122 (60.1)
  Cycle 2 Day 15 6 hours post-dose (ribociclib 400 mg): number analyzed (Participants) | 5
  Cycle 2 Day 15 6 hours post-dose (ribociclib 400 mg) | 72.3 (75.4)
  Cycle 2 Day 15 6 hours post-dose (ribociclib 200 mg): number analyzed (Participants) | 1
  Cycle 2 Day 15 6 hours post-dose (ribociclib 200 mg) | 38.3

13. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from day of participant's informed consent to the day before first dose of study medication.
  On-treatment deaths were collected from start of treatment to 30 days after last dose of treatment or one day before first administration of crossover treatment (for crossover participants), whichever came first Crossover on-treatment deaths were collected from start of crossover treatment up to 30 days after last dose of crossover treatment.
  Post-treatment efficacy/survival follow-up deaths were collected from day 31 after last dose of study treatment to end of study.
  Crossover post-treatment efficacy/survival follow-up deaths were collected from day 31 after last dose of crossover treatment to end of study.
Time Frame: Pre-treatment: Up to 28 days prior to treatment. On-treatment: Up to 82 months. Crossover on-treatment: Up to 3.5 months. Post-treatment efficacy/survival follow-up: Up to 82 months. Crossover post-treatment efficacy/survival follow-up: Up to 1 year
Population: FAS including all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ribociclib + Fulvestrant | Placebo + Fulvestrant
Number analyzed (Participants) | 484 | 242
Participants
  Pre-treatment deaths | 0 | 0
  On-treatment deaths: number analyzed (Participants) | 483 | 241
  On-treatment deaths | 13 | 8
  Crossover on-treatment deaths: number analyzed (Participants) | 0 | 3
  Crossover on-treatment deaths |  | 0
  Post-treatment efficacy/survival deaths: number analyzed (Participants) | 380 | 210
  Post-treatment efficacy/survival deaths | 264 | 153
  Crossover post-treatment efficacy/survival deaths: number analyzed (Participants) | 0 | 1
  Crossover post-treatment efficacy/survival deaths |  | 1
  All deaths | 277 | 162

ADVERSE EVENTS:
Time Frame: On-treatment AEs: from 1st dose to 30 days post-treatment (or start of crossover treatment), up to 82 months. Post-treatment efficacy/survival follow-up deaths: from 31 days post-treatment to end of study, up to 82 months. Crossover on-treatment AEs: from 1st dose to 30 days post-crossover treatment, up to 3.5 months. Crossover post-treatment efficacy/survival follow-up deaths: from 31 days post-crossover treatment to end of study, up to 1 year
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Deaths in the post treatment follow-up period are not considered Adverse Events. The total number at risk in the post treatment includes patients that entered the post treatment follow-up period (post-treatment efficacy and/or survival follow-up). Analysis performed in the safety set including participants who received at least one dose of study treatment
Groups:
- Ribociclib + Fulvestrant (On-treatment): AEs during on-treatment period (up to 30 days after last dose of treatment)
- Ribociclib + Fulvestrant (Post-treatment Efficacy/Survival Follow-up); Placebo + Fulvestrant (Post-treatment Efficacy/Survival Follow-up): Deaths collected in the post- treatment efficacy/survival follow-up period (starting from day 31 post- treatment). No AEs were collected during this period
- Placebo + Fulvestrant (On-treatment): AEs during on-treatment period (up to 30 days after last dose of treatment or one day before first dose of crossover treatment for crossover participants)
- Crossover to Ribociclib + Fulvestrant (Crossover On-treatment): AEs during crossover on-treatment period (from start of crossover treatment up to 30 days after last dose of crossover treatment)
- Crossover to Ribociclib + Fulvestrant (Crossover Post-treatment Efficacy/Survival Follow-up): Deaths collected in the crossover post-treatment efficacy/survival follow-up period (starting from day 31 post-crossover treatment). No AEs were collected during this period
Arm/Group | Ribociclib + Fulvestrant (On-treatment) | Ribociclib + Fulvestrant (Post-treatment Efficacy/Survival Follow-up) | Placebo + Fulvestrant (On-treatment) | Placebo + Fulvestrant (Post-treatment Efficacy/Survival Follow-up) | Crossover to Ribociclib + Fulvestrant (Crossover On-treatment) | Crossover to Ribociclib + Fulvestrant (Crossover Post-treatment Efficacy/Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 13/483 | 264/380 | 8/241 | 153/210 | 0/3 | 1/1
Serious Adverse Events (participants affected / at risk) | 179/483 | 0/0 | 51/241 | 0/0 | 1/3 | 0/0
Other Adverse Events (participants affected / at risk) | 475/483 | 0/0 | 225/241 | 0/0 | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib + Fulvestrant (On-treatment) (N=483) | Ribociclib + Fulvestrant (Post-treatment Efficacy/Survival Follow-up) (N=0) | Placebo + Fulvestrant (On-treatment) (N=241) | Placebo + Fulvestrant (Post-treatment Efficacy/Survival Follow-up) (N=0) | Crossover to Ribociclib + Fulvestrant (Crossover On-treatment) (N=3) | Crossover to Ribociclib + Fulvestrant (Crossover Post-treatment Efficacy/Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 7 | NA | 0 | NA | 0 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | NA | 0 | NA | 0 | NA
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | NA | 0 | NA | 0 | NA
Neutropenia (Blood and lymphatic system disorders) | 7 | NA | 0 | NA | 0 | NA
Pancytopenia (Blood and lymphatic system disorders) | 2 | NA | 0 | NA | 0 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | NA | 0 | NA | 0 | NA
Acute coronary syndrome (Cardiac disorders) | 1 | NA | 0 | NA | 0 | NA
Acute myocardial infarction (Cardiac disorders) | 1 | NA | 1 | NA | 0 | NA
Angina pectoris (Cardiac disorders) | 2 | NA | 0 | NA | 0 | NA
Aortic valve sclerosis (Cardiac disorders) | 1 | NA | 0 | NA | 0 | NA
Atrial fibrillation (Cardiac disorders) | 2 | NA | 0 | NA | 0 | NA
Atrioventricular block second degree (Cardiac disorders) | 1 | NA | 0 | NA | 0 | NA
Bradycardia (Cardiac disorders) | 1 | NA | 0 | NA | 0 | NA
Cardiac failure (Cardiac disorders) | 3 | NA | 0 | NA | 0 | NA
Cardiac failure congestive (Cardiac disorders) | 1 | NA | 0 | NA | 0 | NA
Cardiomyopathy (Cardiac disorders) | 0 | NA | 1 | NA | 0 | NA
Cardiopulmonary failure (Cardiac disorders) | 1 | NA | 0 | NA | 0 | NA
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | NA | 0 | NA | 0 | NA
Myocardial infarction (Cardiac disorders) | 2 | NA | 0 | NA | 0 | NA
Pericardial effusion (Cardiac disorders) | 1 | NA | 0 | NA | 0 | NA
Supraventricular tachycardia (Cardiac disorders) | 1 | NA | 2 | NA | 0 | NA
Tachyarrhythmia (Cardiac disorders) | 1 | NA | 0 | NA | 0 | NA
Tachycardia (Cardiac disorders) | 1 | NA | 1 | NA | 0 | NA
Ventricular arrhythmia (Cardiac disorders) | 1 | NA | 0 | NA | 0 | NA
Vertigo (Ear and labyrinth disorders) | 1 | NA | 0 | NA | 0 | NA
Adrenal insufficiency (Endocrine disorders) | 0 | NA | 1 | NA | 0 | NA
Goitre (Endocrine disorders) | 1 | NA | 0 | NA | 0 | NA
Diplopia (Eye disorders) | 1 | NA | 0 | NA | 0 | NA
Myopia (Eye disorders) | 1 | NA | 0 | NA | 0 | NA
Abdominal distension (Gastrointestinal disorders) | 1 | NA | 0 | NA | 0 | NA
Abdominal pain (Gastrointestinal disorders) | 6 | NA | 1 | NA | 0 | NA
Abdominal pain upper (Gastrointestinal disorders) | 2 | NA | 1 | NA | 0 | NA
Anal incontinence (Gastrointestinal disorders) | 1 | NA | 0 | NA | 0 | NA
Aphthous ulcer (Gastrointestinal disorders) | 1 | NA | 0 | NA | 0 | NA
Ascites (Gastrointestinal disorders) | 1 | NA | 1 | NA | 0 | NA
Colitis (Gastrointestinal disorders) | 1 | NA | 0 | NA | 0 | NA
Constipation (Gastrointestinal disorders) | 4 | NA | 0 | NA | 0 | NA
Diarrhoea (Gastrointestinal disorders) | 2 | NA | 1 | NA | 0 | NA
Dysphagia (Gastrointestinal disorders) | 1 | NA | 0 | NA | 0 | NA
Faecaloma (Gastrointestinal disorders) | 1 | NA | 0 | NA | 0 | NA
Gastric ulcer (Gastrointestinal disorders) | 0 | NA | 1 | NA | 0 | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | NA | 1 | NA | 0 | NA
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | NA | 0 | NA | 0 | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | NA | 0 | NA | 0 | NA
Gingival disorder (Gastrointestinal disorders) | 0 | NA | 1 | NA | 0 | NA
Ileus (Gastrointestinal disorders) | 2 | NA | 0 | NA | 0 | NA
Intestinal obstruction (Gastrointestinal disorders) | 1 | NA | 0 | NA | 0 | NA
Nausea (Gastrointestinal disorders) | 10 | NA | 0 | NA | 0 | NA
Small intestinal obstruction (Gastrointestinal disorders) | 3 | NA | 0 | NA | 0 | NA
Vomiting (Gastrointestinal disorders) | 8 | NA | 1 | NA | 0 | NA
Asthenia (General disorders) | 3 | NA | 0 | NA | 0 | NA
Fatigue (General disorders) | 1 | NA | 0 | NA | 0 | NA
General physical health deterioration (General disorders) | 2 | NA | 2 | NA | 0 | NA
Malaise (General disorders) | 1 | NA | 0 | NA | 0 | NA
Non-cardiac chest pain (General disorders) | 4 | NA | 0 | NA | 0 | NA
Pyrexia (General disorders) | 6 | NA | 1 | NA | 0 | NA
Swelling face (General disorders) | 1 | NA | 0 | NA | 0 | NA
Systemic inflammatory response syndrome (General disorders) | 1 | NA | 0 | NA | 0 | NA
Terminal state (General disorders) | 1 | NA | 0 | NA | 0 | NA
Acute hepatic failure (Hepatobiliary disorders) | 0 | NA | 2 | NA | 0 | NA
Biliary colic (Hepatobiliary disorders) | 0 | NA | 1 | NA | 0 | NA
Cholangitis (Hepatobiliary disorders) | 1 | NA | 0 | NA | 0 | NA
Cholecystitis (Hepatobiliary disorders) | 2 | NA | 0 | NA | 0 | NA
Cholecystitis acute (Hepatobiliary disorders) | 1 | NA | 1 | NA | 0 | NA
Cholelithiasis (Hepatobiliary disorders) | 2 | NA | 1 | NA | 0 | NA
Drug-induced liver injury (Hepatobiliary disorders) | 1 | NA | 1 | NA | 0 | NA
Hepatic cytolysis (Hepatobiliary disorders) | 1 | NA | 0 | NA | 0 | NA
Hepatic failure (Hepatobiliary disorders) | 1 | NA | 0 | NA | 0 | NA
Hepatotoxicity (Hepatobiliary disorders) | 1 | NA | 0 | NA | 0 | NA
Anaphylactic shock (Immune system disorders) | 1 | NA | 0 | NA | 0 | NA
Anal abscess (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Appendicitis (Infections and infestations) | 2 | NA | 0 | NA | 0 | NA
Breast cellulitis (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Bronchitis (Infections and infestations) | 2 | NA | 0 | NA | 0 | NA
COVID-19 (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
COVID-19 pneumonia (Infections and infestations) | 2 | NA | 0 | NA | 0 | NA
Cellulitis (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Clostridium difficile infection (Infections and infestations) | 0 | NA | 1 | NA | 0 | NA
Cystitis (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Diverticulitis (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Erysipelas (Infections and infestations) | 1 | NA | 1 | NA | 0 | NA
Escherichia pyelonephritis (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Gangrene (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Gastroenteritis (Infections and infestations) | 2 | NA | 0 | NA | 0 | NA
Infection (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Influenza (Infections and infestations) | 4 | NA | 1 | NA | 0 | NA
Lower respiratory tract infection (Infections and infestations) | 1 | NA | 1 | NA | 0 | NA
Neutropenic sepsis (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Pneumonia (Infections and infestations) | 13 | NA | 3 | NA | 0 | NA
Pneumonia influenzal (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Postoperative wound infection (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Pyelonephritis (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Respiratory tract infection (Infections and infestations) | 3 | NA | 0 | NA | 0 | NA
Sepsis (Infections and infestations) | 3 | NA | 0 | NA | 0 | NA
Upper respiratory tract infection (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Urinary tract infection (Infections and infestations) | 4 | NA | 2 | NA | 1 | NA
Urosepsis (Infections and infestations) | 2 | NA | 1 | NA | 0 | NA
Viral infection (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Wound infection (Infections and infestations) | 1 | NA | 0 | NA | 0 | NA
Ankle fracture (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Contusion (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Fall (Injury, poisoning and procedural complications) | 5 | NA | 0 | NA | 0 | NA
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Femur fracture (Injury, poisoning and procedural complications) | 2 | NA | 1 | NA | 0 | NA
Foot fracture (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Fracture (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Hip fracture (Injury, poisoning and procedural complications) | 5 | NA | 1 | NA | 0 | NA
Humerus fracture (Injury, poisoning and procedural complications) | 0 | NA | 2 | NA | 0 | NA
Incisional hernia (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | NA | 1 | NA | 0 | NA
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Multiple fractures (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Overdose (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Procedural pain (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Radius fracture (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Rib fracture (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Spinal fracture (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | NA | 1 | NA | 0 | NA
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | NA | 0 | NA | 0 | NA
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | NA | 0 | NA | 0 | NA
Wrist fracture (Injury, poisoning and procedural complications) | 2 | NA | 0 | NA | 0 | NA
Alanine aminotransferase increased (Investigations) | 4 | NA | 0 | NA | 0 | NA
Aspartate aminotransferase increased (Investigations) | 3 | NA | 0 | NA | 0 | NA
Blood alkaline phosphatase increased (Investigations) | 0 | NA | 1 | NA | 0 | NA
Blood creatinine increased (Investigations) | 2 | NA | 0 | NA | 0 | NA
Blood phosphorus decreased (Investigations) | 1 | NA | 0 | NA | 0 | NA
Electrocardiogram QT prolonged (Investigations) | 2 | NA | 1 | NA | 0 | NA
Hepatic enzyme increased (Investigations) | 1 | NA | 0 | NA | 0 | NA
Liver function test abnormal (Investigations) | 1 | NA | 0 | NA | 0 | NA
Liver function test increased (Investigations) | 1 | NA | 0 | NA | 0 | NA
Neutrophil count decreased (Investigations) | 1 | NA | 0 | NA | 0 | NA
White blood cell count decreased (Investigations) | 1 | NA | 0 | NA | 0 | NA
Decreased appetite (Metabolism and nutrition disorders) | 1 | NA | 0 | NA | 0 | NA
Dehydration (Metabolism and nutrition disorders) | 4 | NA | 1 | NA | 0 | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | NA | 2 | NA | 0 | NA
Hypervolaemia (Metabolism and nutrition disorders) | 0 | NA | 1 | NA | 0 | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | NA | 0 | NA | 0 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | NA | 0 | NA | 0 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 2 | NA | 0 | NA | 0 | NA
Hypophagia (Metabolism and nutrition disorders) | 0 | NA | 1 | NA | 0 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | NA | 2 | NA | 0 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 3 | NA | 0 | NA | 0 | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | NA | 2 | NA | 0 | NA
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | NA | 0 | NA | 0 | NA
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | NA | 0 | NA | 0 | NA
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | NA | 0 | NA | 0 | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | NA | 1 | NA | 0 | NA
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | NA | 0 | NA | 0 | NA
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | NA | 1 | NA | 0 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | NA | 1 | NA | 0 | NA
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | NA | 1 | NA | 0 | NA
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | NA | 1 | NA | 0 | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | NA | 1 | NA | 0 | NA
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA | 0 | NA | 0 | NA
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA | 1 | NA | 0 | NA
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | NA | 1 | NA | 0 | NA
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA | 0 | NA | 0 | NA
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | NA | 1 | NA | 0 | NA
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA | 0 | NA | 0 | NA
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | NA | 1 | NA | 0 | NA
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | NA | 1 | NA | 0 | NA
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA | 0 | NA | 0 | NA
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA | 0 | NA | 0 | NA
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA | 0 | NA | 0 | NA
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA | 0 | NA | 0 | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA | 0 | NA | 0 | NA
Aphasia (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA
Carotid artery stenosis (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA
Cerebral haemorrhage (Nervous system disorders) | 1 | NA | 1 | NA | 0 | NA
Cerebral infarction (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA
Cerebral ischaemia (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA
Cerebrovascular accident (Nervous system disorders) | 0 | NA | 1 | NA | 0 | NA
Dizziness (Nervous system disorders) | 4 | NA | 0 | NA | 0 | NA
Dysarthria (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA
Headache (Nervous system disorders) | 2 | NA | 0 | NA | 0 | NA
Hemiparesis (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA
Intercostal neuralgia (Nervous system disorders) | 0 | NA | 1 | NA | 0 | NA
Ischaemic stroke (Nervous system disorders) | 2 | NA | 0 | NA | 0 | NA
Paraesthesia (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA
Presyncope (Nervous system disorders) | 1 | NA | 1 | NA | 0 | NA
Seizure (Nervous system disorders) | 2 | NA | 0 | NA | 0 | NA
Somnolence (Nervous system disorders) | 2 | NA | 0 | NA | 0 | NA
Spinal cord compression (Nervous system disorders) | 2 | NA | 0 | NA | 0 | NA
Syncope (Nervous system disorders) | 2 | NA | 0 | NA | 0 | NA
Transient ischaemic attack (Nervous system disorders) | 1 | NA | 1 | NA | 0 | NA
Trigeminal neuralgia (Nervous system disorders) | 1 | NA | 0 | NA | 0 | NA
Anxiety (Psychiatric disorders) | 1 | NA | 1 | NA | 0 | NA
Confusional state (Psychiatric disorders) | 4 | NA | 0 | NA | 0 | NA
Delirium (Psychiatric disorders) | 1 | NA | 0 | NA | 0 | NA
Disorientation (Psychiatric disorders) | 1 | NA | 0 | NA | 0 | NA
Mental status changes (Psychiatric disorders) | 0 | NA | 1 | NA | 0 | NA
Sleep disorder (Psychiatric disorders) | 1 | NA | 0 | NA | 0 | NA
Acute kidney injury (Renal and urinary disorders) | 6 | NA | 0 | NA | 0 | NA
Bladder hypertrophy (Renal and urinary disorders) | 1 | NA | 0 | NA | 0 | NA
Prerenal failure (Renal and urinary disorders) | 1 | NA | 0 | NA | 0 | NA
Renal failure (Renal and urinary disorders) | 2 | NA | 0 | NA | 0 | NA
Ureteric obstruction (Renal and urinary disorders) | 2 | NA | 0 | NA | 0 | NA
Ureterolithiasis (Renal and urinary disorders) | 1 | NA | 0 | NA | 0 | NA
Urinary tract obstruction (Renal and urinary disorders) | 2 | NA | 0 | NA | 0 | NA
Uterine prolapse (Reproductive system and breast disorders) | 0 | NA | 1 | NA | 0 | NA
Vaginal haematoma (Reproductive system and breast disorders) | 0 | NA | 1 | NA | 0 | NA
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 0 | NA | 0 | NA
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 0 | NA | 0 | NA
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 1 | NA | 0 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 0 | NA | 0 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | NA | 5 | NA | 0 | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 1 | NA | 0 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | NA | 3 | NA | 0 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | NA | 0 | NA | 0 | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | NA | 2 | NA | 0 | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | NA | 3 | NA | 0 | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | NA | 1 | NA | 0 | NA
Rash macular (Skin and subcutaneous tissue disorders) | 1 | NA | 0 | NA | 0 | NA
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | NA | 0 | NA | 0 | NA
Arteriosclerosis (Vascular disorders) | 1 | NA | 0 | NA | 0 | NA
Deep vein thrombosis (Vascular disorders) | 1 | NA | 0 | NA | 0 | NA
Embolism (Vascular disorders) | 1 | NA | 0 | NA | 0 | NA
Hypertension (Vascular disorders) | 1 | NA | 0 | NA | 0 | NA
Hypotension (Vascular disorders) | 2 | NA | 1 | NA | 0 | NA
Ischaemia (Vascular disorders) | 1 | NA | 0 | NA | 0 | NA
Lymphoedema (Vascular disorders) | 1 | NA | 0 | NA | 0 | NA
Shock haemorrhagic (Vascular disorders) | 1 | NA | 0 | NA | 0 | NA
Superior vena cava syndrome (Vascular disorders) | 1 | NA | 0 | NA | 0 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib + Fulvestrant (On-treatment) (N=483) | Ribociclib + Fulvestrant (Post-treatment Efficacy/Survival Follow-up) (N=0) | Placebo + Fulvestrant (On-treatment) (N=241) | Placebo + Fulvestrant (Post-treatment Efficacy/Survival Follow-up) (N=0) | Crossover to Ribociclib + Fulvestrant (Crossover On-treatment) (N=3) | Crossover to Ribociclib + Fulvestrant (Crossover Post-treatment Efficacy/Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 92 | NA | 21 | NA | 2 | NA
Leukopenia (Blood and lymphatic system disorders) | 93 | NA | 1 | NA | 0 | NA
Lymphopenia (Blood and lymphatic system disorders) | 31 | NA | 2 | NA | 0 | NA
Neutropenia (Blood and lymphatic system disorders) | 279 | NA | 6 | NA | 1 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 30 | NA | 5 | NA | 0 | NA
Vertigo (Ear and labyrinth disorders) | 35 | NA | 4 | NA | 0 | NA
Dry eye (Eye disorders) | 28 | NA | 8 | NA | 0 | NA
Lacrimation increased (Eye disorders) | 27 | NA | 2 | NA | 0 | NA
Abdominal pain (Gastrointestinal disorders) | 46 | NA | 18 | NA | 0 | NA
Abdominal pain upper (Gastrointestinal disorders) | 59 | NA | 19 | NA | 0 | NA
Colitis (Gastrointestinal disorders) | 3 | NA | 1 | NA | 1 | NA
Constipation (Gastrointestinal disorders) | 123 | NA | 33 | NA | 0 | NA
Diarrhoea (Gastrointestinal disorders) | 164 | NA | 54 | NA | 1 | NA
Dry mouth (Gastrointestinal disorders) | 27 | NA | 5 | NA | 0 | NA
Dyspepsia (Gastrointestinal disorders) | 56 | NA | 15 | NA | 0 | NA
Dysphagia (Gastrointestinal disorders) | 12 | NA | 3 | NA | 1 | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 25 | NA | 5 | NA | 0 | NA
Nausea (Gastrointestinal disorders) | 226 | NA | 75 | NA | 1 | NA
Stomatitis (Gastrointestinal disorders) | 63 | NA | 13 | NA | 0 | NA
Toothache (Gastrointestinal disorders) | 33 | NA | 5 | NA | 0 | NA
Vomiting (Gastrointestinal disorders) | 135 | NA | 34 | NA | 1 | NA
Asthenia (General disorders) | 74 | NA | 31 | NA | 0 | NA
Fatigue (General disorders) | 164 | NA | 82 | NA | 0 | NA
Influenza like illness (General disorders) | 38 | NA | 17 | NA | 0 | NA
Injection site pain (General disorders) | 25 | NA | 14 | NA | 0 | NA
Non-cardiac chest pain (General disorders) | 25 | NA | 13 | NA | 0 | NA
Oedema peripheral (General disorders) | 70 | NA | 16 | NA | 0 | NA
Pyrexia (General disorders) | 70 | NA | 17 | NA | 0 | NA
Bronchitis (Infections and infestations) | 34 | NA | 12 | NA | 0 | NA
Cystitis (Infections and infestations) | 26 | NA | 9 | NA | 0 | NA
Influenza (Infections and infestations) | 31 | NA | 12 | NA | 0 | NA
Nasopharyngitis (Infections and infestations) | 70 | NA | 34 | NA | 0 | NA
Oral candidiasis (Infections and infestations) | 0 | NA | 0 | NA | 1 | NA
Oral herpes (Infections and infestations) | 11 | NA | 4 | NA | 1 | NA
Pharyngitis (Infections and infestations) | 10 | NA | 5 | NA | 1 | NA
Upper respiratory tract infection (Infections and infestations) | 60 | NA | 19 | NA | 0 | NA
Urinary tract infection (Infections and infestations) | 62 | NA | 29 | NA | 1 | NA
Alanine aminotransferase increased (Investigations) | 77 | NA | 16 | NA | 0 | NA
Amylase increased (Investigations) | 13 | NA | 3 | NA | 1 | NA
Aspartate aminotransferase increased (Investigations) | 70 | NA | 17 | NA | 0 | NA
Blood cholesterol increased (Investigations) | 21 | NA | 14 | NA | 0 | NA
Blood creatinine increased (Investigations) | 44 | NA | 10 | NA | 1 | NA
Electrocardiogram QT prolonged (Investigations) | 30 | NA | 3 | NA | 0 | NA
Gamma-glutamyltransferase increased (Investigations) | 39 | NA | 19 | NA | 0 | NA
Lipase increased (Investigations) | 24 | NA | 14 | NA | 0 | NA
Neutrophil count decreased (Investigations) | 105 | NA | 4 | NA | 0 | NA
Weight decreased (Investigations) | 27 | NA | 12 | NA | 0 | NA
White blood cell count decreased (Investigations) | 66 | NA | 2 | NA | 0 | NA
Decreased appetite (Metabolism and nutrition disorders) | 93 | NA | 32 | NA | 0 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 27 | NA | 11 | NA | 0 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 155 | NA | 91 | NA | 0 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 108 | NA | 46 | NA | 0 | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 49 | NA | 24 | NA | 0 | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 37 | NA | 14 | NA | 0 | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 21 | NA | 23 | NA | 0 | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 27 | NA | 16 | NA | 0 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 49 | NA | 27 | NA | 0 | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 41 | NA | 14 | NA | 0 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 86 | NA | 48 | NA | 0 | NA
Dizziness (Nervous system disorders) | 71 | NA | 22 | NA | 1 | NA
Headache (Nervous system disorders) | 120 | NA | 51 | NA | 0 | NA
Paraesthesia (Nervous system disorders) | 19 | NA | 16 | NA | 0 | NA
Anxiety (Psychiatric disorders) | 34 | NA | 15 | NA | 0 | NA
Depression (Psychiatric disorders) | 38 | NA | 13 | NA | 0 | NA
Insomnia (Psychiatric disorders) | 63 | NA | 30 | NA | 1 | NA
Acute kidney injury (Renal and urinary disorders) | 4 | NA | 1 | NA | 2 | NA
Breast pain (Reproductive system and breast disorders) | 7 | NA | 14 | NA | 0 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 126 | NA | 42 | NA | 0 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 85 | NA | 32 | NA | 0 | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 39 | NA | 17 | NA | 0 | NA
Alopecia (Skin and subcutaneous tissue disorders) | 100 | NA | 12 | NA | 0 | NA
Dry skin (Skin and subcutaneous tissue disorders) | 40 | NA | 8 | NA | 0 | NA
Erythema (Skin and subcutaneous tissue disorders) | 26 | NA | 3 | NA | 0 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 107 | NA | 18 | NA | 0 | NA
Rash (Skin and subcutaneous tissue disorders) | 106 | NA | 19 | NA | 0 | NA
Hot flush (Vascular disorders) | 69 | NA | 40 | NA | 0 | NA
Hypertension (Vascular disorders) | 66 | NA | 26 | NA | 0 | NA
Hypotension (Vascular disorders) | 18 | NA | 6 | NA | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT02422615/Prot_002.pdf
  • Statistical Analysis Plan (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT02422615/SAP_003.pdf